CLINICAL TRIAL: NCT05254574
Title: Sustained Acoustic Medicine for Osteoarthritis Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA-01-2022
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis
Keywords: Continuous ultrasound; Sustained Acoustic Medicine; Musculoskeletal Injuries; Low Intensity Continuous Ultrasound; Pain; Joint Injury; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SAM Ultrasound Device and Diclofenac Patch (Experimental): Patients receive treatment from the wired SAM Ultrasonic Diathermy Device for 4 hours at least 5 days a week for 8 weeks combined with 2.5% diclofenac patch. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Device with 2.5% Diclofenac Patch; Drug: 2.5% Diclofenac Patches

INTERVENTIONS:
Device: Sustained Acoustic Device with 2.5% Diclofenac Patch — Patients apply the SAM Ultrasonic Diathermy Device daily for 1-4 hours of continuous therapeutic ultrasound at 3 megahertz(MHz) frequency and 0.132 Watts/cm@ with 2.5% Diclofenac patches.
  Other Names: ZetrOZ Ultrasound Device; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS DeviceWearable; Long Duration Low-Intensity Device
Drug: 2.5% Diclofenac Patches — Topical pain relief-gel worn for 4 hours at least 5 days a week via SAM patch.

SUMMARY:
The purpose of this study is to compare Sustained Acoustic Medicine treatment to topical pain relief gel for the symptomatic management of osteoarthritis. The study will measure pain and function scores for patients undergoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed mild to moderate knee, shoulder, elbow, ankle, hip, or spine osteoarthritis OA (OARSI atlas grades 1-2) or also referred to as Degenerative Joint Disease (DJD).
* Fulfill the American College of Rheumatology clinical and radiological diagnostic criteria for knee OA
* Are between 35-85 years of age
* Report a frequent pain score between 3-7 (range: 0-10) during the week preceding enrollment
* Report that knee, shoulder, elbow, ankle, hip, or spine pain negatively affects quality of life
* Are willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved treatment provided to the subject at the initiation of the study
* Are deemed appropriate by their physician or by the study site physician to participate.
* Be willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the study device.
* Not use or initiate opioid and/or non-opioid analgesic medications.
* Be willing to discontinue any other interventional treatment modalities on the treatment area during the study period (e.g., transcutaneous electrical nerve stimulation, electronic muscle stimulation, traditional ultrasound).

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device.
* Displays any condition which, in the judgment of the investigator, would make participation in the study unacceptable including, but not limited to, the subject's ability to understand and follow instructions.
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening.
* Is pregnant.
* Is a prisoner.
* Has a pacemaker.
* Has a malignancy in the treatment area.
* Has an active infection, open sores, or wounds in the treatment area.
* Has impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia.
* Has a known neuropathy (disease of the brain or spinal nerves).
* Has a hereditary disposition (tendency) for excessive bleeding (hemorrhage).
* Have knee, shoulder, elbow, ankle, or hip replacement or other surgical intervention, in the affected area in the past 6 months.
* Requires oxygen support
* Has an allergy to aspirin or other NSAIDs
* Have a secondary cause of arthritis (metabolic or inflammatory)

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Units on a Scale (0-10) 0 Being Least, 10 Being Worst Pain From Baseline | Through study completion, average of 8 weeks
  Change in the self described pain units on a scale by patient at baseline and post-
Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Time Frame: Through study completion, average of 8 weeks
  WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index) at baseline and post-treatment to calculate the change in scores. WOMAC was divided into 3 categories: pain, stiffness, function and total score. The pain category consists of five scores from 0 - 4, 0 being no pain 4 is worst pain possible, for a range of 0 - 20 points. The stiffness category consists of two scores from 0 - 4, 0 being no stiffness 10 is worst stiffness possible for a range of 0 - 8 points. The function score consists of 17 scores from 0 - 4, 0 being normal function and 10 is severely limited function, for a range of 0 - 68 points. Total score is the sum of pain, stiffness, and function scores (range of 0 - 96).

SECONDARY OUTCOMES:
Change in Global Rating of Change (GROC) on a Scale (-7 to +7) | Through study completion, average of 24 weeks.
  Subject-reported change in overall pain on a scale, -7 = worst, +7 = best.
Change in the Pain & Sleep Questionnaire (PSQ-3) | Through study completion, average of 24 weeks.
  Subject-reported rating of impact of pain on sleep on a scale from 0 no impact, to 100 greatest impact
Change in Depression Anxiety Stress Scale (DASS21) | Through study completion, average of 24 weeks.
  Subject-reported measures of depression, anxiety, and stress on a scale of 0-3, 0 being not applicable, 1 meaning applicable to some degree, 2 meaning applicable often, and 3 meaning applicable most of the time. Questions are divided into three categories: depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Winkler, Ph.D., Principal Investigator — James A. Haley Veterans Hospital
Locations (1):
- James A Haley Veterans Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madzia A, Agrawal C, Jarit P, Petterson S, Plancher K, Ortiz R. Sustained Acoustic Medicine Combined with A Diclofenac Ultrasound Coupling Patch for the Rapid Symptomatic Relief of Knee Osteoarthritis: Multi-Site Clinical Efficacy Study. Open Orthop J. 2020;14:176-185. doi: 10.2174/1874325002014010176. Epub 2020 Dec 18. PMID 33408796
- [Background] Best TM, Petterson S, Plancher K. Sustained acoustic medicine as a non-surgical and non-opioid knee osteoarthritis treatment option: a health economic cost-effectiveness analysis for symptom management. J Orthop Surg Res. 2020 Oct 19;15(1):481. doi: 10.1186/s13018-020-01987-x. PMID 33076955
- [Background] Draper DO, Klyve D, Ortiz R, Best TM. Effect of low-intensity long-duration ultrasound on the symptomatic relief of knee osteoarthritis: a randomized, placebo-controlled double-blind study. J Orthop Surg Res. 2018 Oct 16;13(1):257. doi: 10.1186/s13018-018-0965-0. PMID 30326947
- [Background] Langer MD, Levine V, Taggart R, Lewis GK, Hernandez L, Ortiz R. Pilot Clinical Studies of Long Duration, Low Intensity Therapeutic Ultrasound for Osteoarthritis. Proc IEEE Annu Northeast Bioeng Conf. 2014 Apr;2014:14789673. doi: 10.1109/NEBEC.2014.6972850. PMID 25788823